CLINICAL TRIAL: NCT00359970
Title: Loperamide Plus Azithromycin More Effectively Treats Travelers' Diarrhea In Mexico Than Azithromycin Alone
Brief Title: Azithromycin, With or Without Loperamide, to Treat Travelers' Diarrhea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Charles D Ericsson, Professor and Dr. and Mrs. Carl V. Vartian Professor in Infectious Diseases, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-02-082
Record Dates: First submitted 2006-08-01; First posted 2006-08-03 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Diarrhea
Keywords: Diarrhea; Travel; Travelers' diarrhea; Azithromycin; Loperamide; Treatment; Antibiotic
MeSH Terms: conditions — Diarrhea | interventions — Azithromycin; Loperamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Azithromycin 500 mg plus Placebo (Active Comparator): a single 500 mg dose of Azitrhomycin at the start of treatment; a single loading dose of placebo at the start of treatment and then a dose of placebo after each loose stool
  Interventions: Drug: Azithromycin 500 mg; Other: Placebo
- Azithromycin 1000 mg plus Placebo (Active Comparator): a single 1000 mg dose of Azitrhomycin at the start of treatment; a single loading dose of placebo at the start of treatment and then a dose of placebo after each loose stool
  Interventions: Drug: Azithromycin 1000 mg; Other: Placebo
- Azithromycin 500 mg plus Loperamide (Experimental): a single 500 mg dose of Azitrhomycin at the start of treatment; a single 4 mg loading dose of Loperamide at the start of treatment and then 2 mg Loperamide after each loose stool
  Interventions: Drug: Azithromycin 500 mg; Drug: Loperamide

INTERVENTIONS:
Drug: Azithromycin 500 mg — A single 500 mg dose at the start of treatment
  Other Names: Zithromax, Zmax
  Arms: Azithromycin 500 mg plus Loperamide; Azithromycin 500 mg plus Placebo
Drug: Azithromycin 1000 mg — A single 1000 mg dose at the start of treatment
  Other Names: Zithromax, Zmax
  Arms: Azithromycin 1000 mg plus Placebo
Drug: Loperamide — A single 4 mg loading dose at the start of treatment and then 2 mg after each loose stool
  Other Names: IModium, Loperamide HCl
  Arms: Azithromycin 500 mg plus Loperamide
Other: Placebo — A single loading dose at the start of treatment and then a dose after each loose stool
  Arms: Azithromycin 1000 mg plus Placebo; Azithromycin 500 mg plus Placebo

SUMMARY:
In a previous study azithromycin proved as efficacious as levofloxacin in the treatment of travelers' diarrhea in Mexico. Because the addition of loperamide to some antibiotics (e.g., trimethoprim-sulfamethoxazole and ofloxacin) has proven more efficacious than antibiotic alone in the treatment of travelers' diarrhea, we decided to study the addition of loperamide to azithromycin.

US adults with acute diarrhea in Guadalajara Mexico were randomized to receive azithromycin in two different doses or loperamide plus azithromycin.

The duration of diarrhea was shorter (11 hours) in the combination-treated group compared to the antibiotic-treated groups (34 hours). The percentage of subjects continuing to pass 6 or more unformed stools in the first 24 hours was less (1.7%) in the combination-treated group than in the antibiotic-treated groups (20%).

We feel loperamide should routinely be added to an antibiotic to optimize treatment of travelers' diarrhea.

DETAILED DESCRIPTION:
Background. The combination of loperamide and trimethoprim-sulfamethoxazole or a fluoroquinolone has proven to be more efficacious than the antimicrobial agent alone in the treatment of travelers' diarrhea. We set out to prove loperamide plus azithromycin was more efficacious that azithromycin alone.

Methods. During the summers of 2002-3, 176 US adults recently arrived in Guadalajara, Mexico were enrolled in a prospective, double-blinded, randomized trial of the treatment of acute diarrhea. Subjects received single doses (1000 mg or 500 mg) of azithromycin or a single 500 mg dose of azithromycin plus loperamide. Subjects gave a pre and post treatment stool sample for analysis and maintained daily diaries of symptoms and passage of stools.

Results. The MIC90 of azithromycin for all E. coli and Shigella was 0.03 and 4 µg/ml with eradication rates in day 5 stools of 88% and 100%, respectively. The duration of diarrhea was significantly (p=0.0002) shorter following treatment with azithromycin plus loperamide (11 h) than with either dose of azithromycin alone (34 h). In the first 24 h the average number of unformed stools passed was 3.4 (azithromycin-alone) and 1.2 (combination) for a significant (p<0.0001) difference of 2.2 unformed stools. This difference equated with 20% of azithromycin-treated subjects continuing to pass 6 or more unformed stools in the first 24 h post treatment compared with only 1.7% of combination-treated subjects.

Conclusions. For the treatment of travelers' diarrhea in an E. coli predominant region of the world a single 500 mg dose of azithromycin appeared as effective as a 1000 mg dose. Loperamide plus 500 mg azithromycin was safe and more effective than either dose of azithromycin. To realize the substantial clinical benefit that accrues to a subset of subjects, we feel loperamide should routinely be used in combination with an antimicrobial agent to treat travelers' diarrhea.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects included men or women, recently arrived in Mexico, at least 18 years of age, who developed acute diarrhea, which was defined as passage of 3 or more unformed stools in the preceding 24 hours accompanied by one or more signs or symptoms of enteric infection (e.g., nausea, vomiting, abdominal cramps, tenesmus, passage of grossly bloody stools or fecal urgency) with a duration of illness of less than or equal to 72 hours.

Exclusion Criteria:

* Exclusion criteria included pregnancy, breast feeding, an unstable medical condition, taking two or more doses of an antidiarrheal medication in the 24 hours before enrollment or any number of doses of symptomatic therapy within 2 hours of enrollment, or receiving an antimicrobial drug with expected activity against enteric bacterial pathogens within 7 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2002-06; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Hours from beginning treatment to passage of last unformed stool | subjects recorded the time and form of all stools passed during a 4 day observation period

SECONDARY OUTCOMES:
Number of unformed stools passed per 24 hour period | 24 hours after treatment
Number of subjects with symptoms of enteric disease per 24 hour period | 24 hours after treatment
  Symptoms of enteric disease include nausea, vomiting, abdominal cramps, gas, urgency, and tenesmus.
Number of treatment failures | 72 hours after treatment
  Treatment failure is defined as persisting ill after 72 hours
Percent of subjects in whom enteropathogen isolated from an enrollment stool sample was eradicated from a day 5 stool | 5 days after treatment
Percent of subjects continuing to pass 3 or more (enrollment criteria) unformed stools in a 24 hour period | 24 hours after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Charles D. Ericsson, MD, Principal Investigator — University of Texas Medical School at Houston
Locations (1):
- University of Texas Enteric Disease Research Clinics, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Background] Adachi JA, Ericsson CD, Jiang ZD, DuPont MW, Martinez-Sandoval F, Knirsch C, DuPont HL. Azithromycin found to be comparable to levofloxacin for the treatment of US travelers with acute diarrhea acquired in Mexico. Clin Infect Dis. 2003 Nov 1;37(9):1165-71. doi: 10.1086/378746. Epub 2003 Sep 30. PMID 14557959
- [Background] Ericsson CD, DuPont HL, Okhuysen PC, Jiang ZD, DuPont MW. Loperamide plus azithromycin more effectively treats travelers' diarrhea in Mexico than azithromycin alone. J Travel Med. 2007 Sep-Oct;14(5):312-9. doi: 10.1111/j.1708-8305.2007.00144.x. PMID 17883462